CLINICAL TRIAL: NCT06945874
Title: Validity and Reliability of the French Translation of the Richards-Campbell Questionnaire for Assessing Sleep in the Intensive Care Unit
Brief Title: Validity and Reliability of the French Translation of the Richards-Campbell Questionnaire
Acronym: French-RCSQ
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/0017/OB; IDRCB : 2025-A00224-45 (Other: ANSM)
Record Dates: First submitted 2025-04-09; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-03

CONDITIONS: Sleep Disorders Not Due to A Substance or Known Physiological Condition
Keywords: sleep disorders in intensive care patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Validation of sleep quality by the Richards-Campbell Sleep Questionnaire (RCSQ) in french version — The RCSQ questionnaire translated into French (RCSQ-F) will be distributed to intensive care patients who meet the inclusion and non-inclusion criteria and who have given their informed consent to participate in the study.
  The questionnaire will be distributed on two occasions: at the first visit and on the day of discharge from intensive care for survivors, or at the latest on the 14th day of hospitalisation.
  Patients' use of the questionnaire will enable internal validation (primary objective) by exploratory factor analysis.

SUMMARY:
The validation of a sleep questionnaire (translated into French from a source questionnaire in English) will provide a reliable and easily administered tool for assessing sleep quality in intensive care, enabling better identification of patients at risk of sleep disorders and other associated complications, in particular ventilatory weaning difficulties.

DETAILED DESCRIPTION:
Sleep disturbance in intensive care is influenced by a number of factors, such as environmental nuisances (noise, light, repeated interruptions), treatments (sedation, analgesia, mechanical ventilation) and the severity of the acute pathology that led to admission. Consequences include alterations to the immune system, neuropsychiatric disorders and impaired functional recovery.

Current management of these disorders remains limited:

* No pharmacological treatment has clearly demonstrated its efficacy on sleep quality in intensive care.
* Interventions aimed at modulating environmental nuisances (reducing noise, reducing light exposure, respecting day/night cycles) have shown limited effects.
* According to the available data, individual devices (eye masks, earplugs) have not significantly improved sleep architecture.

In this context, the Richards-Campbell questionnaire (RCSQ) represents an interesting alternative for subjectively assessing sleep in intensive care patients. This questionnaire, specifically designed for these patients, provides a simple and rapid assessment of sleep disturbances. The validation of a French version of the RCSQ meets a need to standardise assessment practices in France and to gain a better understanding of the factors influencing sleep quality in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Hospitalised in intensive care for at least 24 hours
* Able to understand and answer questionnaires
* Unsedated (discontinued for 24 hours) presenting a Richmond Sedation Agitation Scale score between ≥-2 and ≤ +1
* Fluent in French
* Having given oral consent for participation in the study
* Person affiliated to a social security scheme.

Exclusion Criteria:

* Patient refusal
* Person deprived of liberty by an administrative or judicial decision or protected adult subject (under guardianship or curatorship)
* Patient unable, for whatever reason, to read, understand or answer the questionnaires (visual problems, psychiatric or cognitive problems, etc.)
* Patient already included in the study or another study evaluating sleep

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The RCSQ-F questionnaire will be distributed at the same time as the ISI and Epworth questionnaires to ICU patients who meet the inclusion and non-inclusion criteria and who have given their informed consent to participate in the study.
  The questionnaires will be distributed on two occasions: at the first visit and on the day of discharge from intensive care.
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Validation of the French translation of the Richards-Campbell questionnaire | Visit Inclusion (V1, Day 1) and Visit V2 (Day 14)
  Assessing the internal validity of the French translation of the Richards-Campbell questionnaire for analysing sleep quality in intensive care patients

SECONDARY OUTCOMES:
Inter-rater agreement between patients and nurses | Visit Inclusion (V1, Day 1)
  Evaluation of inter-rater agreement between scores given by patients and nurses. The inter-judge agreement between patient and nurse (first secondary objective) will be evaluated by an intra-class correlation coefficient (single measure, absolute agreement, two-way random) on observations with neither missing data on the patient assessment nor the nurse assessment at the V1 visit.
Convergent validity of the results of the French RCSQ with other questionnaires | Visit Inclusion (V1, Day 1)
  To assess the convergent validity of the results of the French RCSQ with the Epworth scale. This convergent validity (2nd secondary objective) will be assessed by the Pearson correlation coefficient of the overall score of the RCSQ-F with the Epworth on observations with no missing data on these scales at the V1 visit.
Convergent validity of the results of the French RCSQ with other questionnaires | Visit Inclusion (V1, Day 1)
  To assess the convergent validity of the results of the French RCSQ with the ISI scale. This convergent validity (2nd secondary objective) will be assessed by the Pearson correlation coefficient of the overall score of the RCSQ-F with the ISI on observations with no missing data on these scales at the V1 visit.
Divergent validity of results | Visit Inclusion (V1, Day 1)
  Assess the divergent validity of the results by analysing the correlation between the French RCSQ and the HAD scale. This divergent validity will be assessed at V1 by calculating the Pearson correlation coefficient between the total RCSQ-F and the HAD scale: a low correlation coefficient (but not necessarily zero) is desirable: R < 0.30 ideally.
French RCSQ's sensitivity to change | Visit V2 (Day 14)
  To assess the sensitivity to change of the French RCSQ by analysis of subjects with neither missing data at V1 nor missing data at V2 (discharge from intensive care) concerning the RCSQ-F. Sensitivity to change will be assessed by a 95% Student's confidence interval on paired series estimating the difference in standardised means (i.e. divided by the standard deviation at V1) of the total RCSQ-F. The sensitivity to change of each of the RCSQ-F items will be analysed in the same way. The correlation matrix of changes in the items between V1 and V2 will also be calculated, thus verifying the consistency of the evolutionary trends.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Anne MM MELONE, Doctor, Principal Investigator — University Rouen Hospital
Locations (2):
- France (2):
  - University Hospital of Poitiers, Poitiers
  - University Rouen Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.